CLINICAL TRIAL: NCT03332498
Title: A Phase I/II Study of Pembrolizumab in Combination With Ibrutinib for Advanced, Refractory Colorectal Cancers
Brief Title: Pembrolizumab in Combination With Ibrutinib for Advanced, Refractory Colorectal Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19091
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Colon Cancer; Colorectal Cancer; Colorectal Carcinoma; Colon Disease
Keywords: colon; rectum; advanced; refractory
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Colonic Diseases | interventions — pembrolizumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab and Ibrutinib (Experimental): Pembrolizumab intravenously (IV): 200 mg every 3 weeks (Q3W).
  Ibrutinib by mouth (PO): Phase I Dose Escalation at doses of 420 mg daily (cohort 0) and 560 mg daily (cohort 1);. Phase II treatment at Recommended Phase II dose.
  Interventions: Drug: Pembrolizumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Pembrolizumab — 200 milligrams of pembrolizumab will be given through an IV (intravenously) for about thirty minutes. Pembrolizumab is an anti-PD1 that functions by inhibiting checkpoint inhibition and reversing T cell suppression.
  Other Names: Keytruda®
Drug: Ibrutinib — Ibrutinib oral capsules every day starting on cycle 1, day 1. Ibrutinib is primarily a BTK inhibitor which has been approved for the treatment of several hematologic malignancies.
  Other Names: Imbruvica®

SUMMARY:
The purpose of this study is to determine the safety and tolerability, describe the dose-limiting toxicities (DLTs), and determine the maximum tolerated dose (MTD) (or the highest protocol-defined dose level in the absence of establishing an MTD) of ibrutinib in combination with pembrolizumab in participants with advanced, refractory colorectal cancers.

DETAILED DESCRIPTION:
On this study, one treatment cycle equals 21 days. On the first day of each study treatment cycle, 200 milligrams of pembrolizumab will be given through an IV (intravenously) for about thirty minutes. In addition, participants will begin taking the ibrutinib capsules every day starting on cycle 1, day 1. Participants will have a follow-up visit every 3 weeks, on about the first day of each cycle with laboratories drawn to make sure that the study drugs are not causing any side effects. In addition, participants will have a computed tomography (CT) scan every 6 to 7 weeks to determine whether your cancer is getting better or worse.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of colorectal adenocarcinoma.
* Measurable or non-measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Stage IV or recurrent disease is required.
* Participants must have received and progressed through or become intolerant to fluoropyrimidine, irinotecan, oxaliplatin, and bevacizumab. If RAS wild type, participants should have received and progressed or become intolerant to the above as well as cetuximab or panitumumab containing therapies. Prior therapy with Regorafenib and/or TAS 102 is allowed.
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 or 1.
* Estimated life expectancy > 3 months.
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin > 8.0 g/dl
  * Absolute neutrophil count (ANC) > 1,000/mm^3 independent of growth factor support
  * Platelet count > 100,000/mm^3
  * Total bilirubin < 1.5 times upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
  * AST, ALT and Alkaline Phosphatase ≤2.5 times the ULN ( ≤5 x ULN for potential participants with liver involvement)
  * Creatinine clearance ≥ 30 ml/min
* Must not have had chemotherapy, major surgery, monoclonal antibody therapy or experimental therapy within the 21 days prior to the start of ibrutinib administration
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women and surgically sterilized women are not required to undergo a pregnancy test.
* Men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form (ICF) until at least 4 months for both females and males after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Must agree to not donate sperm (males) or eggs (females) during and up to 120 days after the last dose of study treatment.
* Must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure. Must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study requirements.

Exclusion Criteria:

* Active central nervous system (CNS) metastases. If CNS metastases are treated and patients are at neurologic baseline for at least 2 weeks prior to enrollment, they will be eligible but will need a Brain MRI prior to enrollment. Must be off corticosteroids or on a dose of less than 10mg per day.
* Active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* Prior therapy with ibrutinib or other BTK inhibitors.
* Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
* Serologic status reflecting active hepatitis B or C infection. Patients who are hepatitis B core antibody positive and who are antigen negative, will need to have a negative PCR result prior to enrollment. Those who are hepatitis B antigen positive or PCR positive, will be excluded.
* Child Pugh B or C cirrhosis.
* History of severe hypersensitivity reactions to other monoclonal antibodies.
* Substance abuse, medical, psychological or social conditions that may interfere with participation in the study or evaluation of the study results.
* History or concurrent condition of interstitial lung disease of any grade or severely impaired pulmonary function.
* Unresolved toxicity higher than CTCAE grade 1 attributed to any prior therapy or procedure, excluding alopecia.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmia, congestive heart failure, any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or history of myocardial infarction within 6 months prior to first dose with study drug.
* Unable to swallow capsules or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption such as; malabsorption syndrome, resection of the small bowel, or poorly controlled inflammatory bowel disease affecting the small intestine.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon).
* Requires treatment with a strong CYP3A4/5 and/or CYP2D6 inhibitor.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Any illness or medical conditions that are unstable or could jeopardize the safety of the participant and his/her compliance in the study.
* Major surgery or a wound that has not fully healed within 4 weeks of enrollment.
* Vaccinated with live, attenuated vaccines within 4 weeks of enrollment.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Kim DW, Tan E, Zhou JM, Schell MJ, Martinez M, Yu J, Carballido E, Mehta R, Strosberg J, Imanirad I, Kim RD. A phase 1/2 trial of ibrutinib in combination with pembrolizumab in patients with mismatch repair proficient metastatic colorectal cancer. Br J Cancer. 2021 May;124(11):1803-1808. doi: 10.1038/s41416-021-01368-z. Epub 2021 Apr 7. PMID 33828254
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Cohort 0: Dose Escalation (Pembrolizumab and Ibrutinib): Pembrolizumab intravenously (IV): 200 mg every 3 weeks (Q3W). Ibrutinib by mouth (PO): Phase I Dose Escalation at 420 mg daily.
- Phase 1 Cohort 1: Dose Escalation (Pembrolizumab and Ibrutinib): Pembrolizumab intravenously (IV): 200 mg every 3 weeks (Q3W). Ibrutinib by mouth (PO): Phase I Dose Escalation at 560 mg daily
- Phase 2: Treatment at RP2D: Phase 2: Treatment at Recommended Phase 2 Dose (RP2D) - 200 mg Pembrolizumab and 560 mg Ibrutinib
  Pembrolizumab: 200 milligrams of pembrolizumab will be given through an IV (intravenously) for about thirty minutes. Pembrolizumab is an anti-PD1 that functions by inhibiting checkpoint inhibition and reversing T cell suppression.
  Ibrutinib: Ibrutinib oral capsules every day starting on cycle 1, day 1. Ibrutinib is primarily a BTK inhibitor which has been approved for the treatment of several hematologic malignancies.
Period: Overall Study
Arm/Group | Phase 1 Cohort 0: Dose Escalation (Pembrolizumab and Ibrutinib) | Phase 1 Cohort 1: Dose Escalation (Pembrolizumab and Ibrutinib) | Phase 2: Treatment at RP2D
Started | 4 | 4 | 32
Completed | 4 | 4 | 30
Not Completed | 0 | 0 | 2
Not completed — Severe illness prior to Day 1 of treatment | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who consented to study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Cohort 0: Dose Escalation (Pembrolizumab and Ibrutinib) | Phase 1 Cohort 1: Dose Escalation (Pembrolizumab and Ibrutinib) | Phase 2: Treatment at RP2D | Total
Number analyzed (Participants) | 4 | 4 | 32 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 24 | 31
  >=65 years | 1 | 0 | 8 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 15 | 17
  Male | 4 | 2 | 17 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 4 | 29 | 37
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 5 | 5
  White | 4 | 4 | 25 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 32 | 40

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Recommended Phase II Dose (RP2D)
Description: Standard 3+3 Design: The first cohort will enroll a minimum of 3 participants, according to a standard 3+3 design. If 0 out of the first 3 participants in the first cohort experience a dose-limiting toxicity (DLT), then dose escalation will continue as planned. If 1 out of the first 3 participants experience a DLT, then the cohort will be expanded to a total of 6 participants, and if no more than 1 out of 6 participants experiences a DLT in a given dose cohort, dose escalation will continue as planned. If ≥ 2 DLTs are observed in the first dose cohort, the principle investigator will discuss with Janssen on how to proceed. The DLT evaluation period will be defined as the time from the first dose of pembrolizumab and ibrutinib to 42 days after the first dose or if a participant experiences a DLT within this time period.
Time Frame: 42 days post first dose
Population: All participants in Phase 1 portion of study who received at least one dose of study drugs
Measure: Number; unit: mg
Groups:
- Pembrolizumab and Ibrutinib: Pembrolizumab intravenously (IV): 200 mg every 3 weeks (Q3W).
  Ibrutinib by mouth (PO): Phase I Dose Escalation at doses of 420 mg daily (cohort 0) and 560 mg daily (cohort 1)
  Pembrolizumab: 200 milligrams of pembrolizumab will be given through an IV (intravenously) for about thirty minutes. Pembrolizumab is an anti-PD1 that functions by inhibiting checkpoint inhibition and reversing T cell suppression.
  Ibrutinib: Ibrutinib oral capsules every day starting on cycle 1, day 1. Ibrutinib is primarily a BTK inhibitor which has been approved for the treatment of several hematologic malignancies.
Arm/Group | Pembrolizumab and Ibrutinib
Number analyzed (Participants) | 8
mg | 560

2. Primary Outcome: Phase II - Disease Control Rate at 4 Months
Description: Percentage of participants who achieved disease control at 4 months. Disease control rate = Complete Response (CR) + Partial Response (PR) + Stable Disease (SD). Tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and RECIST based immune-related response criteria (irRC).
Time Frame: 4 months
Population: All participants in Phase 2 portion who received at least one dose of study drugs.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Treatment at RP2D
Number analyzed (Participants) | 31
percentage of participants | 13

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Description: Includes only participants who received at least one dose of study drugs.
Arm/Group | Phase 1 Cohort 0: Dose Escalation (Pembrolizumab and Ibrutinib) | Phase 1 Cohort 1: Dose Escalation (Pembrolizumab and Ibrutinib) | Phase 2: Treatment at RP2D
All-Cause Mortality (participants affected / at risk) | 3/4 | 4/4 | 26/32
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/4 | 13/32
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 0: Dose Escalation (Pembrolizumab and Ibrutinib) (N=4) | Phase 1 Cohort 1: Dose Escalation (Pembrolizumab and Ibrutinib) (N=4) | Phase 2: Treatment at RP2D (N=32)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 | 2 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Rib pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain -cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Infections and Infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — brain tumor
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edma limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection-Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Low colostomy output (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 0: Dose Escalation (Pembrolizumab and Ibrutinib) (N=4) | Phase 1 Cohort 1: Dose Escalation (Pembrolizumab and Ibrutinib) (N=4) | Phase 2: Treatment at RP2D (N=32)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 11 (11)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 8 (12)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 9 (9)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (3) | 8 (11)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 5 (5)
CPK increased (Investigations) | 1 (1) | 0 (0) | 3 (4)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 2 (3)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Lymphocyte count decreased (Investigations) | 1 (2) | 1 (1) | 2 (3)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 2 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (2) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight gain (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 2 (2)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 11 (15)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 10 (11)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 8 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 7 (7)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (2) | 1 (1) | 6 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 9 (12)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 8 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 7 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 1 (3) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (4) | 13 (15)
Fever (General disorders) | 1 (1) | 1 (1) | 5 (7)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 5 (5)
General disorders and administration site conditions - Other (General disorders) | 2 (4) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 1 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (6)
Musculoskeletal and connective tissue disorders - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (7) | 3 (22) | 13 (21)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 5 (5)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 7 (10)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Parasthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (2) | 8 (11)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
Hot flashes (Vascular disorders) | 2 (3) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 6 (7)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain -cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications -Other (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified -Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03332498/Prot_SAP_000.pdf